CLINICAL TRIAL: NCT01194648
Title: A Multi-Center Prospective Single Arm Intervention Trial Evaluating Focal Therapy Using High Intensity Focused Ultrasound (Sonablate 500) for Localized Prostate Cancer
Brief Title: Focal Therapy for Prostate Cancer Using HIFU
Acronym: INDEX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000684020; 9945 (Other Grant/Funding Number: NIHR - CPMS ID)
Record Dates: First submitted 2010-09-02; First posted 2010-09-03 (Estimated); Last update posted 2018-04-20 (Actual); Status verified 2018-04

CONDITIONS: Male Erectile Disorder; Prostate Cancer; Therapy-related Toxicity; Urinary Incontinence
Keywords: urinary incontinence; male erectile disorder; therapy-related toxicity; stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer
MeSH Terms: conditions — Erectile Dysfunction; Prostatic Neoplasms; Urinary Incontinence | interventions — High-Intensity Focused Ultrasound Ablation

STUDY DESIGN:
Intervention Model Description: Multi-Centre Prospective Single Arm Intervention Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High Intensity Focused Ultrasound (Other): HIFU, the Intervention
  Interventions: Other: questionnaire administration; Procedure: assessment of therapy complications; Procedure: high-intensity focused ultrasound ablation; Procedure: multiparametric magnetic resonance imaging; Procedure: quality-of-life assessment; Procedure: transperineal prostate biopsy; Procedure: transrectal prostate biopsy

INTERVENTIONS:
Other: questionnaire administration
Procedure: assessment of therapy complications
Procedure: high-intensity focused ultrasound ablation
Procedure: multiparametric magnetic resonance imaging
Procedure: quality-of-life assessment
Procedure: transperineal prostate biopsy
Procedure: transrectal prostate biopsy

SUMMARY:
RATIONALE: Prospective trials using hemi-ablation with high intensity focused ultrasound (HIFU) (Sonablate 500) have demonstrated feasibility, safety, and encouraging functional outcomes and early cancer control with 90% of men achieving trifecta status (no erectile dysfunction, leak-free pad-free continence, cancer control). However, these trials have involved small numbers of patients with men selected for good baseline function. A multi-centre prospective trial within a larger cohort of men that better represents the patient population with prostate cancer (external validity) is required.

DETAILED DESCRIPTION:
Verification of a new therapy as favourable, or equivalent, in outcome to 'standard' care is ideally sought through comparison with another matched control group. Randomised controlled trials (RCTs) offer the best method for minimising systematic bias and revealing the true effect of an intervention or drug. However, RCTs involving treatments of localised prostate cancer have had a historically poor patient uptake, as the reference 'gold' standard of care is not known. In addition, RCTs are expensive to run and involve huge infra-structural support. A number of trials in the USA have been forced to close due to lack of recruitment. The ProStart trial in the UK has also had to close for the same reason. It has been acknowledged by the Food and Drug Agency in the USA that comparative randomized trials will be problematic in this area due to lack of physician and patient equipoise. A randomized trial may be feasible if a pragmatic design is adopted but prior to acceptance of such a design, the number of centres with expertise in this complex intervention (mp-MRI, TTPM, focal HIFU) will need to be increased.

Observational studies are a commonly used alternative to ascertain the effectiveness of a treatment. They are used to observe a treatment effect in a selected group of patients who are presumed to derive benefit from the treatment given. Although methodologically not as robust, and therefore prone to bias, they have some benefits over RCTs. The principal ones are those of enhanced external validity (many patients do not wished to be randomised and therefore refuse participation), and more rapid accrual compared to a randomised design. For this reasons, a single arm medium term follow-up cohort intervention study has been designed. At the time of writing the safety and tolerability aspects of focal therapy by HIFU are known as a result of the Phase I/II studies carried out at UCLH. The results have been presented and exist in the public domain in abstract form but have not yet been published (presented in tables above). These early studies were powered to detect a change in the proportion of men who could obtain an erection sufficient for penetration compared to their status prior to their treatment. The very low event rate for both erectile dysfunction and incontinence indicates that the 'proof of concept' has been demonstrated for focal therapy. Moreover, we can be relatively confident that, in expert hands, focal HIFU is safe. Therefore, a multi-centre study is now required involving a larger group of patients for the following reasons:

1. To evaluate medium term cancer control using histological parameters. Stage two of INDEX will evaluate conversion to radical and systemic therapies and link men to national databases to determine survival in 5 and 10 years.
2. To confirm that focal therapy can lead to low rates of genitourinary and rectal toxicity and minimal impact on quality of life within a large and more representative cohort of patients (greater precision around outcome measures).
3. To demonstrate that the skills (characterization through template prostate mapping and MRI as well as the treatment related skills) acquired by the team at UCLH are indeed transferable to other providers.
4. To calculate costs of care and to model potential cost-effectiveness in comparison to alternative therapies. If this single arm intervention study demonstrates acceptable outcomes to support the findings of the Phase I/II studies, it is anticipated that this preliminary study will lead onto a Phase III evaluation of focal therapy, prior to more widespread use of this technology.

ELIGIBILITY:
1. Histologically proven prostate cancer on trans-rectal or transperineal template prostate biopsies.
2. Prostate biopsy (either TRUS or MRI Targeted or Template):

   * TRUS biopsy: up to burden bilateral disease with maximum 3mm one biopsy on non-dominant side is allowable.
   * MRI targeted and/or Template biopsy within 12 months of entry showing:
   * unilateral disease minimum 3mm of Gleason 3+3 or any Gleason 3+4 or 4+3 but not exceeding Gleason 4+3 overall OR
   * bilateral disease presence of clinically significant cancer on only one side (as determined by histological rules described above) Gleason ≤7 which is concordant with the MRI findings.
3. Stage T1-T2cN0M0 disease, as determined by local guidelines (radiological T3a permitted).
4. Serum PSA </=20ng/ml
5. Life expectancy of >/=10 years.
6. Signed informed consent by patient.
7. An understanding of the English language sufficient to understand

Max Age: 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 354 (Estimated)
Dates: Start 2011-06-29 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Conversion to radical therapy and/or requiring systemic therapy and/or developing metastases and/or dying of prostate cancer | 5 years
  To determine the proportion of men converting to radical therapy and/or requiring systemic therapy and/or developing metastases and/or dying of prostate cancer following focal therapy for localised prostate cancer using HIFU
Conversion to radical therapy and/or requiring systemic therapy and/or developing metastases and/or dying of prostate cancer | 10 years
  To determine the proportion of men converting to radical therapy and/or requiring systemic therapy and/or developing metastases and/or dying of prostate cancer following focal therapy for localised prostate cancer using HIFU

SECONDARY OUTCOMES:
rate of erectile dysfunction | 12 months
  The presence of severe erectile dysfunction at 12 months, as measured by the IIEF-5 questionnaire with or without the use of phosphodiesterase-5 inhibitors, in those with absence of severe erectile dysfunction at baseline
rate of erectile dysfunction | 24 months
  The presence of severe erectile dysfunction at 24 months, as measured by the IIEF-5 questionnaire with or without the use of phosphodiesterase-5 inhibitors, in those with absence of severe erectile dysfunction at baseline
time to return of erectile function | 24 months
  Time to return of erectile function (absence of severe ED on IIEF-15 questionnaire)
rate of urinary incontinence (pad free, leak free and pad-free alone) | 12 months
  Presence of urinary incontinence (any pad usage plus any leakage of urine) as determined by the UCLA-EPIC urinary continence questionnaire, at 12 months, in those men with no urinary incontinence at baseline
rate of urinary incontinence (pad free, leak free and pad-free alone) | 24 months
  Presence of urinary incontinence (any pad usage plus any leakage of urine) as determined by the UCLA-EPIC urinary continence questionnaire, at 24 months, in those men with no urinary incontinence at baseline
time to return of continence (pad free, leak free and pad-free alone) | 24 months
  Time to return of urinary continence (as determined by UCLA-EPIC Urinary domain questionnaire)
rate of loss of ejaculation | 24 months
  rate of loss of ejaculation (as determined by IIEF-15 questionnaire)
rate of loss of orgasm | 24 months
  rate of loss of orgasm (as determined by IIEF-15 questionnaire)
rate of pain during intercourse | 24 months
  rate of pain during intercourse (as determined by IIEF-15 questionnaire)
number of men using phosphodiesterase-5 inhibitors to maintain erectile function | 24 months
  Need for phosphodiesterase-5 inhibitors to maintain erectile function sufficient for penetration up to 24 months
rate of lower urinary tract symptoms | 24 months
  Grading of lower urinary tract symptoms as determined by IPSS scores
rate of bowel toxicity | 24 months
  UCLA-EPIC Bowel Function Questionnaire
anxiety levels | 24 months
  EQ-5D Quality of Life Questionnaire
general health related quality of life | 24 months
  General and prostate health related quality of life measured using EQ-5D Quality of Life questionnaire
proportion of men achieving trifecta status at 12 months | 12months
  Achievement of trifecta status (no severe ED, pad-free leak-free continence, cancer control with absence of clinically significant cancer) at 12 months in those men with good baseline function
proportion of men achieving trifecta status at 24 months | 24 months
  Achievement of trifecta status (no severe ED, pad-free leak-free continence, cancer control with absence of clinically significant cancer) at 24 months in those men with good baseline function
rate of secondary prostate cancer intervention (prostatectomy, radiotherapy, androgen ablation, whole-gland HIFU or cryosurgery) | 24 months
  rate of secondary prostate cancer intervention (prostatectomy, radiotherapy, androgen ablation, whole-gland HIFU or cryosurgery)
risk factors for failure defined as a) presence of any cancer and b) clinically significant cancer at study end | 24 months
  risk factors for failure defined as a) presence of any cancer and b) clinically significant
biochemical (PSA) kinetics including determining the optimal biochemical definition of failure | 24 months
  biochemical (PSA) kinetics including determining the optimal biochemical definition of
describe composite outcomes of failure | 24 months
  describe composite outcomes of failure
Cost-effectiveness | 5years
  To determine the costs of treatment and model potential cost effectiveness using comparative cancer control and functional outcomes at 5 years compared to other cohort trials involving the management of localized prostate cancer
Cost-effectiveness | 10 years
  To determine the costs of treatment and model potential cost effectiveness using comparative cancer control and functional outcomes at 10 years compared to other cohort trials involving the management of localized prostate cancer

CONTACTS AND LOCATIONS:
Overall Officials: Mark Emberton, MD, FRCS, MBBS, Study Chair — University College, London; Hashim Uddinn Ahmed, MD, FRCS, Study Chair — Imperial College London
Locations (1):
- University College London, London, England, United Kingdom